CLINICAL TRIAL: NCT05017064
Title: The Effect of Intraoral Cryotherapy on the Change of Inflammatory Cytokine Levels and Postoperative Endodontic Pain in Teeth With Apical Periodontitis
Brief Title: Intraoral Cryotherapy on Cytokine Levels and Postoperative Endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Cangül Keskin, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 119S397-2
Record Dates: First submitted 2021-08-19; First posted 2021-08-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Apical Periodontitis
Keywords: Endodontics infections
MeSH Terms: conditions — Periapical Periodontitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy group (Experimental): An intraoral ice pack will be placed on the mucosal groove during root canal treatment.
  Interventions: Device: Cryotherapy group
- Control group (Placebo Comparator): No ice pack will be used.
  Interventions: Other: Control group

INTERVENTIONS:
Device: Cryotherapy group — The use of intraoral ice pack during root canal treatment
  Arms: Cryotherapy group
Other: Control group — No cryotherapy will be used
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effects of intraoral cryotherapy on the inflammatory cytokine levels during root canal treatment and postoperative pain intensity and incidence. Mandibular premolar teeth of 30 patients diagnosed with asymptomatic apical periodontitis will be included to the study for this purpose. The experimental protocols consist clinical and laboratory phases. In clinical phase, procedures of cryotherapy and control groups will be applied in 2-visit-root canal treatment. The samples, which were collected during root canal treatment, will be subjected to enzyme-linked immunosorbent assay (ELISA) analysis in laboratory. Levels of interleukin and inflammatory destructive enzymes will be determined in collected samples. During the analysis of visual analogue scale scores, the correlation between the changes of the cytokine and proteolytic enzyme levels and presence and intensity of pain will be evaluated.

DETAILED DESCRIPTION:
Cryotherapy is the reduction of the temperature of living tissues for therapeutic purposes. The temperature decrease that will occur as a result of cryotherapy depends on the degree of the applied tissue and agent, the application time, and the thermal permeability of the tissues and the agent . With the application of cryotherapy in human tissues, it is aimed to reduce the temperature of the host cells and control pain.

There is limited data on the use of cryotherapy, which is widely used in medicine, in the field of operative dentistry. It is frequently used after surgical procedures such as cryotherapy, periodontal surgery, tooth extraction and implant application, but its first use in endodontics is to extend the cold saline solution of during root canal treatment. It has been described in laboratory studies that it reduces the external temperature of the root by applying it with apical negative pressure irrigation system for 5 minutes following the procedures. Following this in vitro study, the efficacy of different cryotherapy protocols in reducing pain after root canal treatment was reported by all of the few clinical studies. Studies reported that after endodontic treatment of teeth with symptomatic apical periodontitis, pain severity decreased after cryotherapy application and the frequency of postoperative painkiller use of patients decreased. It was reported that cryotherapy application in endodontic treatments of teeth with symptomatic irreversible pulpitis with vital pulp reduced postoperative pain severity. A laboratory study performed on extracted teeth reported that cryotherapy application reduces the vertical fracture strength of the roots, however, comprehensive laboratory and clinical studies evaluating the various physical properties of the teeth are required in order to make definitive interpretations concerning the clinic and to create a consensus.It has not been fully revealed how and by what mechanism intra-canal cryotherapy applications reduce pain. When cold is applied, a decrease in blood flow occurs in living tissues; It has been shown that neural receptors are inhibited in skin and subcutaneous tissues. Clinical studies report that cold therapy reduces acute musculoskeletal pain, muscle spasms, connective tissue strains, nerve conduction time, and hemorrhage. Cryotherapy restricts the inflammatory reactions that occur in the damaged area by causing vasoconstriction and inhibition of cellular metabolism. Vasoconstriction thus causes a decrease in edema and blockage of nerve endings with the decrease in temperature leads to a decrease in pain. Although decreasing body temperature also decreases peripheral nerve conduction, when it falls below 15 ° C, nerve conduction is completely deactivated. Tissue damage that may result from secondary hypoxia is also minimized by slowing down cell metabolism. The activities and amounts of destructive enzymes in the tissue are reduced. The analgesic effect of cryotherapy is achieved by a combination of reducing the chemical mediators of pain and slowing down neural pain signals. In addition, a 50% slowdown in metabolism has a positive effect on oxygen diffusion in damaged tissues. How intra-canal cryotherapy reduces postoperative endodontic pain has not been fully elucidated yet. When the effects of cryotherapy applications on damaged muscle and connective tissues are interpreted, a decrease in the amount of inflammatory cytokines is expected in a region where cryotherapy is applied. The amounts of inflammatory cytokines and destructive enzymes in periradicular tissues were not evaluated after intra-canal cryotherapy.

Intra-canal cryotherapy stands out as a simple, economical and non-toxic pain control technique, although it eliminates the side effects that may be caused by drugs by reducing the use of painkillers after the procedure. It is a technique that should be applied rather than an alternative, especially for patients who are recommended to avoid painkiller use (drug allergy, geriatric population). It consists of washing the root canals with cold saline solution for 5 minutes, which can be easily adapted to the endodontic treatment routine. This procedure can be applied with negative pressure irrigation systems or endodontic irrigation needles used in routine irrigation. It is a more practical and controlled procedure than applying an ice pack inside or outside the mouth after the procedure, and it will be applied by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy,
* Signing the consent form,
* Having a single-rooted tooth diagnosed with asymptomatic apical periodontitis, -No pre-made restoration, no root canal treatment, no fractures or cracks in the tooth

Exclusion Criteria:

* Not being systemically healthy,
* Not giving consent to the study,
* Presence of cracks, fractures, restorations in the relevant tooth,
* History of Raynaud's phenomenon

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
1.Change of proinflammatory cytokine levels | 12 months
  The samples are collected from periapical exudate at the end of the first and second visit of root canal treatment. The samples are analyzed with high sensitive ELISA method and change of proinflammatory cytokines from first and second visit will be evaluated in ng/ml or pg/ml.
2.Levels of postoperative pain | 12 months
  The intensity of postoperative pain will be evaluated with visual analogue scale, which is a 10 cm line representing a continuum of pain levels between "no pain" on the left side and "most severe pain" on the right side between 0 and 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University Dp. Endodontics, Faculty of Dentistry, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No